CLINICAL TRIAL: NCT06209125
Title: Early Correction of Skeletal Class II Division I by the Hybrid Aesthetic Functional Appliances
Brief Title: Evaluation of Skeletal and Dental Effect of the New Hybrid Aesthetic Functional Appliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sohaila Adnan, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sohaila; IRB approval number (Other: A05051021)
Record Dates: First submitted 2024-01-07; First posted 2024-01-17 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): use new device for treatment of class II malocclusion
  Interventions: Device: hybrid aesthetic functional appliance

INTERVENTIONS:
Device: hybrid aesthetic functional appliance — treatment of class II division one malocclusion

SUMMARY:
use new hybrid aesthetic functional appliance for treatment of class II div 1 malocclusion.

DETAILED DESCRIPTION:
The Sample:

The sample size was calculated using PASS 15 Power Analysis and Sample Size Software (2017). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass.

A sample size of 16 data pairs achieves 80.3% power to reject the null hypothesis of zero effect size when the population effect size is 1.00 and the significance level (alpha) is 0.050 using a two-sided paired t-test.

The ten patients will be selected from the outpatient clinic of the Orthodontic Department, Faculty of Dentistry, Mansoura University.

The parents of each patient will be informed regarding the study and will sign written consent before starting the treatment.

Records:

1. Photographs:

   1. Extra-oral (frontal -lateral -frontal with a smile).
   2. Intra-oral (frontal -lateral - occlusal).
2. Radiographs:

   1. Cephalometric.
   2. Panorama.
   3. Hand wrist radiographs.
3. Upper and lower orthodontic casts.

Appliance construction:

* After taking the upper and lower impressions; a construction wax bite will be done, and the mandible will be positioned anteriorly to achieve an edge-to-edge relationship parallel to the functional occlusal plane. Single-step advancement of the mandible will be achieved If the overjet ranges between (3-4 mm) or segmental advancement if it is larger than 5 mm using the Exactobite.
* HAF appliance will be constructed It is of double plate design, consisting of thermoplastic and acrylic parts The upper component is a vacuum-formed plate, made of transparent hard-elastic polyethylene sheet with 2 mm thickness, equipped with an acrylic advancement bar positioned in the anterior midpalatal region.

Similarly, the lower plate is constructed by thermoplastic material of the same width covering the six anterior teeth.

An acrylic guidance surface is placed over the plastic coverage on the lingual surfaces of lower incisors and canines, aimed to fit the upper bar.

Two-sided arms are extended from the acrylic resin body up to second molars adapted to the morphology of the lingual vestibule.

To obtain optimal shape matching of the opposing attachments, the working casts are mounted on a semi-adjustable articulator to contact in an end-to-end relationship.

Posterior teeth are intentionally exposed to facilitate eruption and leveling of a deep curve of Spee.

White-colored acrylic resin is used for the fabrication of acrylic parts to enhance esthetics.

Using a special plier, buttons are formed at the cervical third of upper and lower dental midlines to enable night-time wear of vertical elastics, or light-cured composite resin combined with appropriate transparent matrices can be used for button construction.

* The patients will be instructed to:

  * use the HAF appliance for 12-14 hours per day.
  * Maintain good oral hygiene, and brush your teeth after each meal.
  * Attain an orthodontic clinic every three weeks.
  * Use elastics at night.
* When the overjet is corrected; the upper part is served shortly as the anterior bite plane.

ELIGIBILITY:
Inclusion Criteria:

* Age included is the mixed dentition stage ( 6 -12 y )
* skeletal Class II division 1.
* Overjet more than 4 mm.

Exclusion Criteria:

* Previous orthodontic treatment.
* Bad oral hygiene.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Early correction of skeletal classII division I by the hybrid aesthetic functional appliances (HAF) | one year
  early treatment of class II division 1 malocclusion using HAF appliance and evaluate the skeletal and dental effect of new appliance by take cephalogram before and after treatments

CONTACTS AND LOCATIONS:
Overall Officials: sohaila ad ahmed, master, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No